CLINICAL TRIAL: NCT00448487
Title: Prospective Observational Study to Asses the Incidence of CVD Complications in Diabetic Patients Pre-stratified by Haptoglobin Phenotype From the I CARE Registry
Brief Title: Haptoglobin Phenotype and Cardiovascular Complications in Diabetic Patients
Acronym: ICARER
Status: Completed | Type: Observational
Sponsor: Dr. Shany Blum (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor-Investigator, Dr. Shany Blum, Adjunct assistant professor, Technion, Israel Institute of Technology
Organization: Technion, Israel Institute of Technology (Other)
Other Study IDs: KL-2007
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes; Cardiovascular Disease; Myocardial Infarction
Keywords: Diabetes; Cardiovascular Disease; Haptoglobin
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
3054 diabetic patients were screened for Haptoglobin Phenotype as part of the ICARE study (NCT00220831) and composite the I CARE Registry, 1434 Hp 2-2 patients were treated as part of the I CARE study with vitamin E vs. Placebo, this study was recently terminated due to significant differences between the groups and data was sent to publication. All other patients were passively followed since April 2005 for cardiovascular events. We have decided to continue and follow these patients till end of December 2007 to determine the incidence of CVD in theses patients which are pre stratified by Haptoglobin Phenotype.

DETAILED DESCRIPTION:
3054 diabetic patients from Clalit Medical Services were screened for Haptoglobin Phenotype as part of the ICARE study (NCT00220831) and composite the I CARE registry, 1434 Hp 2-2 patients were treated as part of the I CARE study with vitamin E vs. Placebo, this study was recently terminated due to significant differences between the groups and data was sent to publication.

During the follow up period of the I CARE study all 3054 registry patients were followed in a passive way, which means that the patients were not called for follow up visits but the reports for CVD events were centrally collected from patient's Hospital admission summaries. Admission summaries were collected using the computerized systems of the Clalit Health Services assuring that when ever a patient in the registry is hospitalized for what ever reason the study coordination them would be aware of that and receive the admission summary. An events adjudication committee adjudicated each event in a blinded fashion to determine the nature of the events.

1434 patients who were treated by vitamin E or placebo in the I CARE study were also followed by follow-up telephone calls.

once I CARE study was officially terminated we have decided to continue and follow the whole 3054 registry patients in the same manner to complete a nearly 3 year follow up to determine in a prospective manner the incidence of CVD events in Diabetic patients which were pre-stratified by Haptoglobin type.

ELIGIBILITY:
These are the same patients as in I CARE registry so the criteria are the same as was for I CARE study Recruitment phase.

Inclusion Criteria:

* Diabetic patients aged 55 and above

Exclusion Criteria:

* Patient who takes antioxidant treatment will be asked to stop, or can't be included in the study
* Patients who had a CVD incident (MI, Stroke, TIA), Unstable angina pectoris, Uncontrolled HTN, will have to wait a month after stabilization to be included in the study
* Allergy to Vitamin E

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients recruited from primary care clinics. all are diabetic patients 55 years old or older.
Sampling Method: Probability Sample
Enrollment: 3054 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
same as in ICARE: composite major CVD outcomes (non fatal MI, Stroke and CVD death) | Continuously till end of June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Shany Blum, M.D. M.Sc., Principal Investigator — Technion, Israel Institute of Technology; Uzi Milman, M.D., Principal Investigator — Clalit Health Services; Chen Shapira, M.D., Principal Investigator — Clalit Health Services; Andrew P Levy, M.D. Ph.D., Principal Investigator — Technion, Israel Institute of Technology
Locations (1):
- Clalit Health Services, Haifa and Western Galilee District, Haifa, Israel